CLINICAL TRIAL: NCT06830226
Title: The Effect of Domperidone on the Macronutrient and Energy Content of Breastmilk of Mothers With Preterm Delivery, Using a Human Milk Mid-infrared Spectroscopy Analyzer: a Study Protocol
Brief Title: Domperidone on the Composition of Preterm Breastmilk Using a Human Milk Mid-infrared Spectroscopy Analyzer
Acronym: DompMilk
Status: Enrolling by invitation | Type: Observational
Sponsor: Centro Hospitalar de Lisboa Central (Other)
Responsible Party: Sponsor
Other Study IDs: CHULC.CI.633.2025
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-02

CONDITIONS: Insufficient Breast Milk Syndrome; Premature Birth
Keywords: breast milk; domperidone; energy; galactagogue; human milk analyzer; macronutrients; mid-infrared spectroscopy; premature birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Biospecimen Retention: Samples Without DNA — Breast milk from mothers who have delivered prematurely
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test group: Breast milk macronutrient and energy content assessed by mid-infrared spectroscopy method
  Interventions: Dietary Supplement: Test group
- Reference group: Breast milk macronutrient and energy content assessed by Kjeldahl and Röse-Gottlib methods
  Interventions: Dietary Supplement: Reference group

INTERVENTIONS:
Dietary Supplement: Test group — In this group the Miris Human Milk analyzer will be used, consisting of a real-time mid-infrared technology that directly measures the concentration of protein, fat and carbohydrate, and calculates the energy content based on direct measurements.
  Groups: Test group
Dietary Supplement: Reference group — In this group the Kjeldahl method will be used to assess total nitrogen concentration, the Röse-Gottlib method to assess fat concentration, and energy and carbohydrate concentration will be calculated by differences. Kjeldahl and the Röse-Gottlib are considered reference methods
  Groups: Reference group

SUMMARY:
Maintaining milk production in lactating mothers who have delivered prematurely can be a challenge. In these cases, domperidone has been the most commonly used pharmacologic galactagogue. There are several studies on the effect of this drug on the volume of milk produced, but data on its effect on the macronutrient and energy content is scarce. The mid-infrared spectroscopy is a convenient validated method to assess human milk macronutrient and energy content because it requires little training for its operation and a small volume of milk. This study aims to determine the effect of domperidone on the macronutrient and energy content of milk from women who have delivered prematurely, and to compare the results obtained with those reported using reference methods for this analysis.

DETAILED DESCRIPTION:
Study design: This is a single-center observational study based on a convenience cohort of lactating women who have delivered before 37 weeks gestation.

Study period: A consecutive recruitment of participants will be scheduled over 12 months (from February 2, 2025), according to the availability of the observer (M.C.) in charge of the analysis of breast milk in the unit, performed weekly on a routine basis, in order to be fortified if necessary (Cardoso 2023).

Settings: Neonatal Intensive Care Unit (NICU) and Human Milk Bank at Maternidade Dr. Alfredo da Costa, Unidade Local de Saúde São José, Lisbon.

Product to be analyzed: breast milk Demographic variables: Retrieved demographic and clinical variables will include participant age and gestational age at delivery, reported body weight and height closer to the beginning of pregnancy, type of delivery (vaginal or cesarean), parity, pathological conditions during pregnancy (hypertension, pre-eclampsia, gestational diabetes, and intrauterine growth restriction), date of initiation of domperidone, whether it was prescribed by a health professional or on their own initiative, domperidone dosage, and days of lactation at the time of breast milk analyses.

Method of collection and analysis of breast milk: as described in previous studies (Macedo MHNP 2018, Cardoso 2021), mothers will be asked to save milk collected through 24 hours in the same container, in order to minimize daily variability of breast milk composition. The breast milk macronutrient and energy content will be analyzed using the Miris Human Milk analyzer (Miris AB, Uppsala, Sweden).

Measured breast milk macronutrient and energy content: The breast milk macronutrient and energy content will be analyzed using the Miris® Human Milk analyzer (Miris AB, Uppsala, Sweden) following the milk collection and analysis procedures described (Czosnykowska-Łukacka 2018, Macedo MHNP 2018, Cardoso 2021). Before each use, the analyzer will be calibrated using the standard calibration solution (Quan 2020). The breast milk composition will be expressed in densities: Kcal/dL of energy and g/dL of fat, total and true protein, carbohydrates, and ashes (Macedo MHNP 2018, Cardoso 2021).

According to the Unit's routine, the milk of mothers of preterm infants, particularly very preterm infants, is analyzed weekly to assess the need for fortification (Cardoso 2023).

Within-subject differences in the macronutrient and energy milk content will be determined by comparing the value of each parameter (total and true protein, total fat, total carbohydrates and energy) in the last measurement before starting domperidone (M0) with the respective value 14 days after starting (M14).

Estimate of sample size: The study sample size was calculated to detect an effect size of 0.35 between pairs of breastmilk content in total protein, with a significance level of 0.05, and an 80% power; thus, a required sample of 81 infants (67 participants more 20% for drop out) was estimated.

Statistical Analyses Mean of breastmilk macronutrient content will be compared by paired-t test for normal distributed differences or Wilcoxon test if non-normal distributed differences.

ELIGIBILITY:
Inclusion Criteria:

* Lactating women who have delivered prematurely using domperidone as a galactagogue, who will consent to participate, and who are not taking other substances or medications acting as galactagogues

Exclusion Criteria:

* Lactating women do not agree to participate
* Lactating women use domperidone not as a galactagogue
* Lactating women currently or previously taking other substances or medications acting as galactagogues
* Lactating women taking medications that may alter the effect (such as ranitidine) or interact with domperidone (such as haloperidol)
* Lactating women who have the diagnosis of mastitis
* Lactating women with debilitating chronic illness

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Lactating women who have delivered prematurely using domperidone as a galactagogue
Sampling Method: Non-Probability Sample
Enrollment: 81 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
True protein content | Between the last assessment before starting domperidone and the assessment 14 days after starting domperidone. The difference value between 14 days after domperidone and before starting it, expressed as percentage of the value before starting domperidone
  Within-subject difference of breastmilk content in true protein (protein with nutritional value)

SECONDARY OUTCOMES:
Total protein | Between the last assessment before starting domperidone and the assessment 14 days after starting domperidone. The difference value between 14 days after domperidone and before starting it, expressed as percentage of the value before starting domperidone
  Within-subject difference of breastmilk content in total protein
Fat | Between the last assessment before starting domperidone and the assessment 14 days after starting domperidone. The difference value between 14 days after domperidone and before starting it, expressed as percentage of the value before starting domperidone
  Within-subject difference of breastmilk content in fat
Carbohydrate | Between the last assessment before starting domperidone and the assessment 14 days after starting domperidone. The difference value between 14 days after domperidone and before starting it, expressed as percentage of the value before starting domperidone
  Within-subject difference of breastmilk content in carbohydrate
Total energy content | Between the last assessment before starting domperidone and the assessment 14 days after starting domperidone. The difference value between 14 days after domperidone and before starting it, expressed as percentage of the value before starting domperidone
  Within-subject difference of breastmilk content in total energy
Percentage differences for total protein | Between the last assessment before starting domperidone and the assessment 14 days after starting domperidone. The difference value between 14 days after domperidone and before starting it, expressed as percentage of the value before starting domperidone
  The mean of the percentage differences for total protein obtained in the test group will be compared with the correspondent value obtained in the reference group.
Percentage differences for true protein | Between the last assessment before starting domperidone and the assessment 14 days after starting domperidone. The difference value between 14 days after domperidone and before starting it, expressed as percentage of the value before starting domperidone
  7The mean of the percentage differences for true protein obtained in the test group will be compared with the correspondent value obtained in the reference group
Percentage differences for fat | Between the last assessment before starting domperidone and the assessment 14 days after starting domperidone. The difference value between 14 days after domperidone and before starting it, expressed as percentage of the value before starting domperidone
  The mean of the percentage differences for fat obtained in the test group will be compared with the correspondent value obtained in the reference group
Percentage differences for carbohydrate | Between the last assessment before starting domperidone and the assessment 14 days after starting domperidone. The difference value between 14 days after domperidone and before starting it, expressed as percentage of the value before starting domperidone
  The mean of the percentage differences for carbohydrate obtained in the test group will be compared with the correspondent value obtained in the reference group
Percentage differences for total energy | Between the last assessment before starting domperidone and the assessment 14 days after starting domperidone. The difference value between 14 days after domperidone and before starting it, expressed as percentage of the value before starting domperidone
  The mean of the percentage differences for total energy obtained in the test group will be compared with the correspondent value obtained in the reference group

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Virella, MD, MSc, Study Chair — Unidade Local de Saúde São José
Locations (1):
- Unidade Local de Saúde São José, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Czosnykowska-Lukacka M, Krolak-Olejnik B, Orczyk-Pawilowicz M. Breast Milk Macronutrient Components in Prolonged Lactation. Nutrients. 2018 Dec 3;10(12):1893. doi: 10.3390/nu10121893. PMID 30513944
- [Result] Cardoso M, Virella D, Papoila AL, Alves M, Macedo I, E Silva D, Pereira-da-Silva L. Individualized Fortification Based on Measured Macronutrient Content of Human Milk Improves Growth and Body Composition in Infants Born Less than 33 Weeks: A Mixed-Cohort Study. Nutrients. 2023 Mar 22;15(6):1533. doi: 10.3390/nu15061533. PMID 36986263